CLINICAL TRIAL: NCT01790061
Title: Efficacy, Durability and Safety of Standardized Fecal Microbiota Transplantation in Patients With Moderate to Severe Ulcerative Colitis
Brief Title: Standardized Fecal Microbiota Transplantation for Ulcerative Colitis
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Collaborators: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Faming Zhang, Associate professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMT-CN-121123
Record Dates: First submitted 2013-02-09; First posted 2013-02-13 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Bacteria; Microbiota; Fecal Microbiota Transplantation; Inflammatory Bowel Disease; Ulcerative Colitis
Keywords: Gut bacteria; Gut flora; Bacteriotherapy; Fecal Microbiota Transplantation; Inflammatory bowel disease; Ulcerative colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standardized FMT (Experimental): endoscopy Tubing Once or repeat
  Interventions: Procedure: Standardized FMT
- Traditional treatments (Experimental): Oral Tubing
  Interventions: Drug: Traditional treatments

INTERVENTIONS:
Procedure: Standardized FMT — Fecal microbiota transplantation by gastroscopy administration of fresh or frozen bacteria from healthy donor to the mid-gut or whole colon
  Other Names: Fecal Microbiota Transplantation; Fecal Microbiota Therapy; fecal transplantation
  Arms: Standardized FMT
Drug: Traditional treatments — Medications
  Other Names: Traditional treatments according to associated guidelines
  Arms: Traditional treatments

SUMMARY:
The gut microbiota is considered to constitute a "microbial organ" which has pivotal roles in the intestinal diseases and body's metabolism. Evidence from animal and human studies strongly supports the link between intestinal bacteria and inflammatory bowel diseases (IBD). Dozens of studies reported its efficacy in treatment of severe Clostridium difficile colitis. Preliminary studies using FMT for Ulcerative Colitis (UC), Crohn's diseases, irritable bowel syndrome (IBS) and constipation have also met with some success. This is an initial step into investigating the potential efficacy of standardized fecal bacteriotherapy through mid-gut (at least below duodenal papilla) for UC, the investigators propose to determine the efficiency and safety of FMT in a series of 500 patients with moderate to severe UC (Montreal classification).

DETAILED DESCRIPTION:
The present clinical trial aims to re-establish a gut functionality state of intestinal microbiota through FMT as a therapy for UC. Investigators established a standard bacteria isolation from donated fresh stool in lab. Then the bacteria is transplanted to mid-gut through regular gastroscope. Patients in this study will assigned to receive FMT(s) or traditional treatments according to associated guidelines and follow-up for long term. All data were recorded in China Microbiota Transplantation System.

ELIGIBILITY:
Inclusion Criteria:

Patients who had been diagnosed with UC through a combination of typical clinical symptoms, endoscopy, and histological criteria for at least 3 months, and patients who failed to achieve satisfactory efficacy for UC from the previous therapies.

Exclusion Criteria:

Patients were excluded if accompanied by other severe diseases, including other intestinal diseases (e.g., Clostridioides difficile infection), malignant neoplasm, cardiopulmonary failure, and serious liver and kidney disease, refused to complete the follow-up, and underwent FMT or WMT before.

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2013-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of FMT | On year
  The efficacy and durability of clinical remission (days) after Fecal Microbiota Transplantation procedure.Defined as Montreal score S0 (clinical remission)

SECONDARY OUTCOMES:
Adverse events | Ten years
  Number and severity of adverse events
sleep quality evaluated by the Pittsburgh Sleep Quality Index (PSQI) | before FMT, 1 month and 12 weeks after FMT
  Sleep quality was assessed by the Pittsburgh Sleep Quality Index (PSQI), which consisted of 19 items divided into seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.Each component received a value from 0 to 3 and the total scores ranged from 0 to 21, with higher scores indicating poorer sleep quality. Poor sleep quality was defined as total PSQI scores > 5.
sleep quality evaluated by the Insomnia Severity Index (ISI) | before FMT, 1 month and 12 weeks after FMT
  Insomnia Severity Index (ISI) was used to evaluate the severity of insomnia, which was composed of 7 items. Each item scored from 0-4, with a total score ranging from 0 to 28. High scores indicated poorer sleep quality. ISI ≥ 8 was set as a subthreshold to clinical insomnia.
anxiety and depression evaluated by the Hospital Anxiety and Depression Scale (HADS) | before FMT, 1 month and 12 weeks after FMT
  It had 14 items, 7 each for depression (HADS-D) and anxiety (HADS-A). The total scores ranged from 0 to 21 for HADS-D or HADS-A, with higher score indicating more severe depression or anxiety symptoms. A HADS-A or HADS-D score ≥ 8 was identified as a diagnostic threshold for anxiety or depression in this study.
fatigue evaluated by the Functional Assessment of Chronic Illness Therapy fatigue subscale (FACIT-F) | before FMT, 1 month and 12 weeks after FMT
  FACIT-F was composed of 13 questions, each with a score of 0-4. Total score ranged from 0 to 52, with lower score suggesting greater fatigue. Fatigue remission was defined as FACIT-F score > 40 after FMT and an increase in the FACIT-F score ≥ 4 indicated fatigue improvement according to the previous study.

CONTACTS AND LOCATIONS:
Overall Officials: Huijie Zhang, MD,PhD, Study Chair — The Second Afiliated Hospital of Nanjing Medical University
Locations (1):
- Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Borody TJ, Khoruts A. Fecal microbiota transplantation and emerging applications. Nat Rev Gastroenterol Hepatol. 2011 Dec 20;9(2):88-96. doi: 10.1038/nrgastro.2011.244. PMID 22183182
- [Background] Aroniadis OC, Brandt LJ. Fecal microbiota transplantation: past, present and future. Curr Opin Gastroenterol. 2013 Jan;29(1):79-84. doi: 10.1097/MOG.0b013e32835a4b3e. PMID 23041678
- [Background] Zhang F, Luo W, Shi Y, Fan Z, Ji G. Should we standardize the 1,700-year-old fecal microbiota transplantation? Am J Gastroenterol. 2012 Nov;107(11):1755; author reply p.1755-6. doi: 10.1038/ajg.2012.251. No abstract available. PMID 23160295
- [Background] Bennet JD, Brinkman M. Treatment of ulcerative colitis by implantation of normal colonic flora. Lancet. 1989 Jan 21;1(8630):164. doi: 10.1016/s0140-6736(89)91183-5. No abstract available. PMID 2563083
- [Derived] Lu G, Zhang S, Wang R, Wu X, Chen Y, Wen Q, Cui B, Zhang F, Li P. Fecal microbiota transplantation improves bile acid malabsorption in patients with inflammatory bowel disease: results of microbiota and metabolites from two cohort studies. BMC Med. 2025 Sep 1;23(1):511. doi: 10.1186/s12916-025-04353-y. PMID 40890737
- [Derived] Zhang S, Lu G, Wang W, Li Q, Wang R, Zhang Z, Wu X, Liang C, Liu Y, Li P, Wen Q, Cui B, Zhang F. A predictive machine-learning model for clinical decision-making in washed microbiota transplantation on ulcerative colitis. Comput Struct Biotechnol J. 2024 Aug 24;24:583-592. doi: 10.1016/j.csbj.2024.08.021. eCollection 2024 Dec. PMID 39281978
- [Derived] Li Q, Liu Y, Zhang Z, Zhang S, Ding X, Zhang F. Washed Microbiota Transplantation Improves the Sleep Quality in Patients with Inflammatory Bowel Disease. Nat Sci Sleep. 2024 Aug 2;16:1141-1152. doi: 10.2147/NSS.S460882. eCollection 2024. PMID 39109266
- [Derived] Zhang T, Li P, Wu X, Lu G, Marcella C, Ji X, Ji G, Zhang F. Alterations of Akkermansia muciniphila in the inflammatory bowel disease patients with washed microbiota transplantation. Appl Microbiol Biotechnol. 2020 Dec;104(23):10203-10215. doi: 10.1007/s00253-020-10948-7. Epub 2020 Oct 16. PMID 33064186
- [Derived] Li Q, Ding X, Liu K, Marcella C, Liu X, Zhang T, Liu Y, Li P, Xiang L, Cui B, Wang J, Bai J, Zhang F. Fecal Microbiota Transplantation for Ulcerative Colitis: The Optimum Timing and Gut Microbiota as Predictors for Long-Term Clinical Outcomes. Clin Transl Gastroenterol. 2020 Aug;11(8):e00224. doi: 10.14309/ctg.0000000000000224. PMID 32955197
- [Derived] Li Q, Zhang T, Ding X, Xiang L, Cui B, Buch H, Zhang F. Enhancing patient adherence to fecal microbiota transplantation maintains the long-term clinical effects in ulcerative colitis. Eur J Gastroenterol Hepatol. 2020 Aug;32(8):955-962. doi: 10.1097/MEG.0000000000001725. PMID 32282545
- [Derived] Ding X, Li Q, Li P, Zhang T, Cui B, Ji G, Lu X, Zhang F. Long-Term Safety and Efficacy of Fecal Microbiota Transplant in Active Ulcerative Colitis. Drug Saf. 2019 Jul;42(7):869-880. doi: 10.1007/s40264-019-00809-2. PMID 30972640
- [Derived] Cui B, Li P, Xu L, Zhao Y, Wang H, Peng Z, Xu H, Xiang J, He Z, Zhang T, Nie Y, Wu K, Fan D, Ji G, Zhang F. Step-up fecal microbiota transplantation strategy: a pilot study for steroid-dependent ulcerative colitis. J Transl Med. 2015 Sep 12;13:298. doi: 10.1186/s12967-015-0646-2. PMID 26363929
- See also: Fecal microbiota transplantation — http://www.ncbi.nlm.nih.gov/pubmed